CLINICAL TRIAL: NCT02037451
Title: The Effects of Auditory Cueing on Rhythmic Movement and Cortical Excitability in Patients With Parkinson's Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chang Gung University (Other)
Responsible Party: Principal Investigator, Ya-Ju Chang, Profesor, Chang Gung University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 102-3809A3
Record Dates: First submitted 2014-01-14; First posted 2014-01-16 (Estimated); Last update posted 2014-01-16 (Estimated); Status verified 2014-01

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's disease; Auditory Cueing
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- intervention group (Experimental): intervention group which receive auditory cueing while performing movement
  Interventions: Procedure: rhythmic auditory stimulation
- Control group (No Intervention): control group which performing movement after listen to required movement rhythm.

INTERVENTIONS:
Procedure: rhythmic auditory stimulation — Participants perform the finger tapping at the same time give rhythmic auditory stimulation ,and need to execute tapping with auditory stimulation.
  Arms: intervention group

SUMMARY:
Parkinson's disease (PD) is a progressive degenerative disease of central nervous systems deficit. The clinical symptoms of Parkinson's disease include the following motor tasks: difficult in initiating movement, performing rhythmic movement or serial movement, the ability of learning motor movement is also affected. The primary treatment for Parkinson's disease is medical treatment; surgery is used if in need. Rehabilitation such as physical therapy, which aims to improve patient's quality of life and functions, is a non-invasive treatment and value for PD patients. Auditory cue is a technique that widely applied on training patients with Parkinson's disease, and some researches revealed that auditory cueing could improve motor performance. However, the mechanism under this treatment technique is still unknown.

This study is to investigate the effect of auditory cueing on rhythmic finger movement in patients with Parkinson's disease. To investigate the mechanism under auditory cueing, neurophysiological data such as motor cortex excitability and blood flow in cortical cortex will be obtained by using Transcranial magnetic stimulation (TMS) and near infrared spectroscopy (NIRS).

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Parkinson disease

Exclusion Criteria:

* Clinical diagnosis of other neurological diseases
* Dementia
* Been diagnosed with any mental illness
* History of seizures
* Brain trauma
* Body with a pacemaker or other electrical stimulator
* Pregnancy

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2013-08; Primary Completion 2014-08 (Estimated); Study Completion 2014-08 (Estimated)

PRIMARY OUTCOMES:
Finger Tapping | Baseline,45-60 minutes.
  Record pre-test and post-test change.
Motor evoked potential | Baseline,45-60 minute
  Use single-pulse TMS to assess Motor evoked potential change.
Intracortical inhibition & Intracortical facilitation | Baseline,45-60 minutes
  Use paired-pulse TMS to record pre-test and post-test change.
Blood oxygen dependent level | Baseline, in experiment,45-60 minutes
  Use Near-infrared spectroscopy to record pre-test, in experiment, and post-test change.

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung University, Taoyuan District, Taiwan